CLINICAL TRIAL: NCT00211757
Title: Divalproex Sodium vs. Placebo in Childhood/Adolescent Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-0294; 1R21NS043979 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2018-12-06 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Autism
Keywords: autism; aggression; irritability; divalproex sodium
MeSH Terms: conditions — Autistic Disorder; Aggression | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Placebo (Placebo Comparator): Subjects in this arm will receive a placebo comparative to the study drug divalproex sodium.
  Interventions: Drug: Placebo
- Divalproex Sodium (Experimental): Subjects will receive the study drug, divalproex sodium.
  Interventions: Drug: Divalproex sodium

INTERVENTIONS:
Drug: Divalproex sodium — Study drug.
  Arms: Divalproex Sodium
Drug: Placebo — Placebo comparator.
  Arms: Placebo

SUMMARY:
The study is designed to assess the efficacy of treatment with divalproex sodium (DS) vs. placebo in childhood/adolescent autism fulfilling DSM-IV and Autism Diagnostic Interview (ADI) criteria. Currently, there are no FDA-approved treatments for this disorder, although behavioral and educational therapies and a variety of medications may play a role in the management of some autistic symptoms.

DETAILED DESCRIPTION:
This study compares divalproex sodium and placebo in the treatment of autistic disorder. Twenty six child or adolescent outpatients, with age ranges from 5-17, will be randomized into a 12-week double-blind, placebo-controlled parallel treatment study. During the 12 weeks, patients will be monitored by the treating psychiatrist and assessed by an independent evaluator (IE). The IE will perform study assessments while remaining blind to medication regimens (including possible tapering) as well as any side effects. Study assessments will be administered at designated time points

ELIGIBILITY:
Meets DSM-IV, ADI, and ADOS criteria for autistic disorder

Age 5-17.

Outpatients

Parent/legal guardian signing informed consent, and assent documented for patient with demonstrated capacity to provide it.

Sexually active females of childbearing potential must use an acceptable method of birth control (oral contraceptive medications [the administration of which must be supervised by a parent or guardian], IUD, depot medication or tubal ligation) and have a negative serum pregnancy test prior to entry into the study.

Subject scores at least "4" (moderately ill) on the Clinical Global Impression-Severity Scale for Autistic Disorder (CGI-AD).

Subject meets the following criteria at pre-study diagnostic assessment and baseline assessment: OAS-M 13 or ABC-Irritability Subscale 18 (raw scores).

Subjects with history of seizures, who have been seizure-free for 6 months on a stable dose of anticonvulsant medication other than divalproex sodium or related formulations (e.g., depakene). Non-medicated subjects with a history of seizures who have been seizure-free for 6 months. Subjects with abnormal EEG but no clinical seizures.

State exclusion criteria for enrollment in study:

Subjects who are pregnant or nursing mothers. Sexually active women of childbearing potential who are not using adequate birth control measures (detailed above in inclusion criteria).

Subjects with overall adaptive behavior scores below the age of two years on the Vineland Adaptive Behavior Rating Scale.

Subjects with active or unstable epilepsy.

Subjects with any of the following past or present mental disorders: schizophrenia, schizoaffective disorder or organic mental disorders.

Subjects who are a serious suicidal risk.

Subjects with clinically significant or unstable medical illness that would contraindicate participation in the study, including hematopoietic or cardiovascular disease, pancreatitis, liver toxicity, and polycystic ovary syndrome.

Subjects reporting history of encephalitis, phenylketonuria, tuberous sclerosis, fragile X syndrome, anoxia during birth, pica, neurofibromatosis, hypomelanosis of Ito, hypothyroidism, Duchenne muscular dystrophy, and maternal rubella.

Patients with history of the following:

gastrointestinal, liver, or kidney, or other known conditions which will presently interfere presently with the absorption, distribution, metabolism, or excretion of drugs; cerebrovascular disease or brain trauma; clinically significant unstable endocrine disorder, such as hypo- or hyperthyroidism; recent history or presence of any form of malignancy

Treatment within the previous 30 days with any drug known to a well-defined potential for toxicity to a major organ

Subjects with clinically significant abnormalities in laboratory tests or physical exam.

Subjects likely to require ECT or any other psychotropic medication during the study, unless otherwise permitted.

Subjects unable to tolerate taper from psychoactive medication if necessary.

Subjects with a history of hypersensitivity or severe side effects associated with the use of divalproex sodium, or other an ineffective prior therapeutic trial of divalproex sodium (serum levels within range of 50-100 ug/ml for 6 weeks).

Subjects who have received any of the following interventions within the prescribed period before starting treatment:

investigational drugs within the previous 30 days; depot neuroleptic medication; psychotropic drugs not permitted for concurrent use in the study within the previous seven days; fluoxetine within the previous five weeks.

Subjects who have begun any new alternative non-medication treatments, such as diet, vitamins, and psychosocial therapy, within the previous three months.

Subjects with any organic or systemic disease or patients who require a therapeutic intervention, not otherwise specified, which would confound the evaluation of the safety of the study medication.

Subjects who reside in a remote geographical area who do not have regular access to transportation to the clinical facility.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2002-09; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Divalproex Sodium
Started | 11 | 16
Completed | 10 | 14
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lack of Efficacy | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Divalporex Sodium: Subjects will receive the study drug, divalproex sodium.
  Divalproex sodium: Study drug.
- Total: Total of all reporting groups
Arm/Group | Placebo | Divalporex Sodium | Total
Number analyzed (Participants) | 11 | 16 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 16 | 27
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 10 | 13 | 23
Diagnosis [Count of Participants; unit: Participants] — Subjects were either diagnosed with Autistic Disorder or Asperger's syndrome
  Participants
    Autistic Disorder | 9 | 14 | 23
    Asperger's Syndrome | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Improvement on the Clinical Global Impression
Description: The CGI-I is a 7-point improvement scale. Ratings of 1 or 2 (responders) indicate a substantial reduction in symptoms. A rating of 3 (minimally improved) on the CGI is defined as a slight symptomatic improvement that is not deemed clinically significant; patients with such an improvement were not considered responders. Two versions of this test were used, one focused on irritability (primary outcome measure) and a general version CGI-I-autism focused on all symptoms including core symptom domains. The CGI-I irritability took into consideration the scores from the ABC-Irritability subscale, the OAS-M aggression and irritability subscales and information from open-ended questioning related to the degree of interference, nature, and range of behavioral problems at school and at home
Time Frame: Baseline to end of study (week 15)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Divalproex Sodium
Number analyzed (Participants) | 11 | 16
Participants | 1 | 10

2. Primary Outcome: Change in Aberrant Behaviors as Measured by the Aberrant Behavior Checklist Scores
Description: The Aberrant Behavior Checklist is designed to objectively identify five behavior sub scales through observation by the primary caregiver: irritability, lethargy, stereotypy, hyperactivity, and inappropriate speech. The ABC was filled out by parents on a scale from 0-3 for each category. (0 being not a problem, 3 being severe problem). Scores from all sub scales were added (scoring 0-45 for Irritability subscale, 0-48 for Lethargy subscale, 0-21 for stereotypy scale, 0-48 for hyperactivity sub-scale, and 0-12 for inappropriate speech sub-scale) to obtain an overall score with a an overall scoring range of 0-174. Higher scores were indicative of worsening symptoms.
Time Frame: Baseline and End of Study (week 15)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Placebo: Subjects in this arm will receive a placebo comparative to the study drug divalporex sodium.
  Placebo: Placebo comparator.
Arm/Group | Placebo | Divalproex Sodium
Number analyzed (Participants) | 11 | 16
score on a scale
  baseline | 22 (7.81) | 20.3 (7.36)
  Week 15 | 14.5 (6.67) | 17.7 (7.94)

ADVERSE EVENTS:
Time Frame: 6 weeks on treatment
Arm/Group | Placebo | Divalproex Sodium
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/16
Other Adverse Events (participants affected / at risk) | 8/11 | 7/16
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=11) | Divalproex Sodium (N=16)
Insomnia (General disorders) | 2 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Weight gian (Metabolism and nutrition disorders) | 1 | 1
headache (General disorders) | 0 | 1
polyuria (General disorders) | 0 | 2
agitation (General disorders) | 1 | 2
Infection (Immune system disorders) | 3 | 2
Hypersomnolence (General disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No